CLINICAL TRIAL: NCT02541279
Title: Effectiveness of a Group Intervention for the Treatment of Shoulder Pathologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Hospital Universitario San Juan de Alicante (Other)
Responsible Party: Principal Investigator, María Isabel Tomás-Rodríguez, PT, PT MSC, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/324
Record Dates: First submitted 2015-07-31; First posted 2015-09-04 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group received 6 sessions of shoulder exercises controlled by a physiotherapist.
  Interventions: Procedure: Physiotherapy exercises guideline
- Control (Active Comparator): The control group received a paper explaining the same exercises which were performed by the intervention group. This group made the exercises at home.
  Interventions: Procedure: Physiotherapy exercises guideline

INTERVENTIONS:
Procedure: Physiotherapy exercises guideline — Exercises controlled by a physiotherapist.

SUMMARY:
The investigators determined the effectiveness of a group intervention for the treatment of shoulder pathologies.

DETAILED DESCRIPTION:
The investigators performed a two-armed prospective clinical trial study, analyzing a sample formed by 76 patients with shoulder pain. The patients were allocated to one group randomly (intervention or control group). The data was obtained in the San Juan de Alicante Hospital between November 2014 and July 2015.

ELIGIBILITY:
Inclusion Criteria:

-Patients who came to the Rehabilitation Service of the San Juan de Alicante Hospital between November 2014 and July 2015 with one of the diagnosed diseases indicated in the 726.10 ICD-9-CM code (nontraumatic rotator cuff tear, bursitis, tendinitis, and medical diagnostics impingement syndrome of any severity depending stadiums Neer (1990) unilateral or bilateral joint balance with free or minimally limited internal rotation).

Exclusion Criteria:

* Patients who cannot perform the exercises correctly (example: psychiatry disorders)
* Patients with Shoulder surgery
* Patients whose shoulder pain is above 7 according VAS pain.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Constant Murley Test | before/after intervention ( 6 weeks)
  This test assesses daily activities.

SECONDARY OUTCOMES:
Quick-DASH Test | before/after intervention ( 6 weeks)
  This test assesses functional limitation in upper limb musculoskeletal disorders.
Pain NRS (numeric rating scale) | before/after intervention ( 6 weeks)
  Instruct the patient to choose a number from 0 to 10 that best describes their current pain. 0 would mean 'No pain' and 10 would mean 'Worst possible pain'
Measurement of the average force | before/after intervention ( 6 weeks)
  Average force: Measurement was assessed in newtons

CONTACTS AND LOCATIONS:
Overall Officials: M Rosario Asensio Garcia, Phd, Principal Investigator — Universidad Miguel Hernández de Elche Alicante Spain
Locations (1):
- Miguel Hernández de Elche, San Juan, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bervoets DC, Luijsterburg PA, Alessie JJ, Buijs MJ, Verhagen AP. Massage therapy has short-term benefits for people with common musculoskeletal disorders compared to no treatment: a systematic review. J Physiother. 2015 Jul;61(3):106-16. doi: 10.1016/j.jphys.2015.05.018. Epub 2015 Jun 17. PMID 26093806
- [Background] Senbursa G, Baltaci G, Atay A. Comparison of conservative treatment with and without manual physical therapy for patients with shoulder impingement syndrome: a prospective, randomized clinical trial. Knee Surg Sports Traumatol Arthrosc. 2007 Jul;15(7):915-21. doi: 10.1007/s00167-007-0288-x. Epub 2007 Feb 28. PMID 17333123
- [Background] Bankes MJ, Emery RJ. An evaluation of the Constant-Murley shoulder assessment. J Bone Joint Surg Br. 1997 Jul;79(4):696. No abstract available. PMID 9250771
- [Background] Littlewood C, Bateman M, Brown K, Bury J, Mawson S, May S, Walters SJ. A self-managed single exercise programme versus usual physiotherapy treatment for rotator cuff tendinopathy: a randomised controlled trial (the SELF study). Clin Rehabil. 2016 Jul;30(7):686-96. doi: 10.1177/0269215515593784. Epub 2015 Jul 9. PMID 26160149
- [Background] Page MJ, McKenzie JE, Green SE, Beaton DE, Jain NB, Lenza M, Verhagen AP, Surace S, Deitch J, Buchbinder R. Core domain and outcome measurement sets for shoulder pain trials are needed: systematic review of physical therapy trials. J Clin Epidemiol. 2015 Nov;68(11):1270-81. doi: 10.1016/j.jclinepi.2015.06.006. Epub 2015 Jun 16. PMID 26092288
- [Derived] Asensio-Garcia MDR, Bernabeu-Casas RC, Palazon-Bru A, Tomas-Rodriguez MI, Nouni-Garcia R. Effectiveness of a Group Physiotherapy Intervention in Nontraumatic, Inoperable Painful Shoulder: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2018 Feb;97(2):110-115. doi: 10.1097/PHM.0000000000000817. PMID 28857770